CLINICAL TRIAL: NCT03473834
Title: Responses of Modified Exercise Programme on Improvement of Axial Rigidity and Turning Dysfunction in Individuals With Parkinson's Disease
Brief Title: Modified Exercise Programme in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MU-CIRB 2017/181.1210
Record Dates: First submitted 2018-03-07; First posted 2018-03-22 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Exercise; Rigidity; Turning
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Muscle Rigidity | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Only patients with PD who meet the inclusion and exclusion criteria will be invited to participate in the study. All participants will be assessed for daily activity and motor skill using the Unified Parkinson's Disease Rating Scale (UPDRS). At pre- and post- assessments, eye movement and turning characteristics will be assessed using xIMU sensors and EOG.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified exercise programme (Experimental): Modified exercise program is the intervention for the exercise group that they will be received this programm over 1 month.
  Interventions: Other: Modified exercise programme; Behavioral: Medication
- Parkinson's disease Medication (Active Comparator): Medication is the standard treatment for individuals with Parkinson's disease. Therefore, the control group will be received the medication only.
  Interventions: Behavioral: Medication

INTERVENTIONS:
Other: Modified exercise programme — The exercise will be modified from the standardized exercise program (Schenkman, 1998) includes a series of exercises based on the concept that muscle length and coordination.
  Arms: Modified exercise programme
Behavioral: Medication — The control group will be received the normal medication from their doctor.

SUMMARY:
A feasibility study using measures of turning function derived from Inertial Measurement Unit sensory before, and after, a modified exercise programme approach.

DETAILED DESCRIPTION:
Participants will be patients diagnosed as having idiopathic PD by a neurologist. Patients will be recruited from the Movement Disorder Clinic, Division of Neurology, Faculty of Medicine Siriraj Hospital, Mahidol University, Thailand. Participants will be classified into two groups; the treatment and the control groups. All participants will be asked to sign an informed consent form approved by the ethical committee of Mahidol University Institutional Review Board, Mahidol University, Thailand. Only patients with PD who meet the inclusion and exclusion criteria will be invited to participate in the study. All participants will be assessed for daily activity and motor skill using the Unified Parkinson's Disease Rating Scale (UPDRS). At pre- and post- assessments, eye movement and turning characteristics will be assessed using Inertial Measurement Unit sensors and Electroocculography (EOG). The treatment group will receive a rehabilitation program by the physiotherapist. The rehabilitation sessions will take place at the Faculty of Physical Therapy, Mahidol University, Thailand. The control group will receive a diary for recording their daily activities during the duration of participation in this study. In addition, the researcher will phone participants once per week to remind then to maintain their diary records.

Data Processing & Analysis: this study will be used the outcome measures and processing data in MATLAB.

Statistical analysis: Kolmogorov Smirnov Goodness of Fit Test will be used to test the data distribution. If the data are normal or non-normal distribution, data comparisons will be tested as the following;

* Normal distribution: Mixed model ANOVA will be used to compare outcome measures between pre- and post- and between the treatment and the control groups
* Non-normal distribution: The Mann-Whitney U test will be used to compare outcome measures between the treatment and control groups. Wilcoxon Signed-Rank test will be used to compare outcome measures between pre- and post- assessments within group.

ELIGIBILITY:
Inclusion Criteria:

* Presenting clinical diagnosis of Parkinson's disease stage 2 to 3 by modified Hoehn and Yahr Scale assessment
* Age ranges from 50-75 years
* Having stable PD medication usage at least 1 month
* No wearing-off phenomenon
* Able to walk independently without using any assistive device
* Able to follow commands and instruction

Exclusion Criteria:

* Presenting clinical diagnosis of dementia
* Having other neurological, cardiopulmonary, or lower extremities musculoskeletal problems which influence the test performance.
* Having high blood pressure [more than 140/90 mmHg]
* Having hemodialysis
* Having visual problems which cannot be adjusted by the lens or glasses

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Reorientation onset of body segment | 5 months
  Previous research has shown that turning in healthy adults is a whole-body coordinated process characterized by a top-down sequence of body segments reorientation starting with the eyes and head followed by the trunk and ending with the feet (Hollands, Ziavra, & Bronstein, 2004; Mak et al., 2008). However, Lohnes and Earhart (2011) provided evidence that impaired turn performance in PD patients could be partially explained by eye movement deficits, affecting eye, head and body coordination (Lohnes & Earhart, 2011).
Functional Reach test | 5 months
  To assess clinical balance
Fall Efficacy Score (FES-I) | 5 months
  FES-I is a questionnaire to assess fear of falling (31). There is 16-item which developed by the Prevention of Falls Network Europe group (ProFaNE) to augment content covered by the original 10-item Fall Efficacy Score (FES). Participants will be asked to rate 16 items of questionnaire on a four-point Likert scale which is their concerns about the possibility of falling when performing 16 activities. A total score is 64 score, a higher score indicates a greater fear of falling.
Unified Parkinson's Disease Rating Scale (UPDRS) | 5 months
  The Unified Parkinson's Disease Rating Scale, abbreviated UPDRS is a scoring system widely used for the clinical evaluation of Parkinson's disease (PD). Its 42 items are evaluated by interview and clinical observation. Clinicians and researchers alike use the UPDRS and the motor section in particular to follow the progression of a person's Parkinson's disease. Scientific researchers use it to measure benefits from a given therapy in a more unified and accepted rating system. Neurologists also use it in clinical practice to follow the progression of their patients' symptoms in a more objective manner.
  A total of 199 points are possible (199 represents the worst disability and 0 no disability).
Body Mass Index (BMI) | 5 months
  weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Borge Scale | 5 months
  To monitor and quantify individual's perceptions of effort during exercise. The Borge scale is used to measure the intensity of your exercise. The Borge scale runs from 0 - 10. The numbers below relate to phrases used to rate how easy or difficult you find an activity. For example, 0 (nothing at all) would be how you feel when sitting in a chair; 10 (very, very heavy) is how you feel at the end of an exercise stress test or after a very difficult activity.

CONTACTS AND LOCATIONS:
Overall Officials: Fuengfa Khobkhun, Principal Investigator — Mahidol University
Locations (1):
- College of Sports Science and Technology, Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The research is not finished yet when we finish it, we will decide it again.